CLINICAL TRIAL: NCT06744556
Title: HAV Versus DAV/IAV Induction Regimen in Elderly Patients With Acute Myeloid Leukemia Suitable for Intensive Chemotherapy: a Multicenter, Randomized, Controlled Clinical Trial
Brief Title: HAV Versus DAV/IAV Induction Regimen in Elderly Patients With AML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024095
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-11

CONDITIONS: AML
Keywords: Elderly Patients
MeSH Terms: interventions — Daunorubicin; venetoclax; Cytarabine; Azacitidine; Homoharringtonine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAV/IAV (Active Comparator): Induction therapy:
  Ara-C 100mg/m2/d, d1-5 Daunorubicin 60mg/m2/d, d1-2 or Idarubicin 10mg/m2/d, d1-2 Venetoclax 100mg d3, 200mg d4,400mg d5-11 If the treatment achieves CR/CRi/CRh, proceed directly to consolidation therapy.
  If the treatment does not achieve CR/CRi/CRh, enter the second induction phase with a different treatment regimen.
  Second Induction Phase:
  For patients with FLT3 or IDH1 mutations, targeted therapy can be chosen. If there is no FLT3 or IDH1 mutation or the patient is unwilling to use FLT3 or IDH1 inhibitors, switch to the HAV induction regimen.
  Consolidation therapy:
  1. intermediate-dose Ara-C (ID-Ara-C): 2 cycles are used. Ara-C 1 g/m2/q12h on days 1, 3, and 5 (for patients aged 60-70 years) or Ara-C 500 mg/m2/q12h on days 1, 3, and 5 (for patients aged 70 years or older)
  Maintenance therapy:
  VA regimen: 6 courses Azacitidine 75 mg/m2/d on days 1-5, Venetoclax 400 mg on days 1-7.
  Interventions: Drug: daunorubicin; Drug: Venetoclax; Drug: cytarabine; Drug: azacitidine; Drug: Idarubicin
- HAV (Experimental): Induction Therapy:
  Ara-C 100mg/m2/d, d1-5 HHT 2mg/m2/d, d1-5 Venetoclax 100mg d3, 200mg d4,400mg d5-11 If CR/CRi/CRh is achieved, proceed directly to consolidation therapy. If the treatment does not reach CR/CRi/CRh, enter the second induction phase with a different treatment regimen.
  Second course:
  For patients with FLT3 or IDH1 mutations, the corresponding targeted therapy can be selected, as before.
  For patients without FLT3 or IDH1 mutations or those who do not want to use FLT3 or IDH1 inhibitors, the DAV/IAV induction regimen is changed.
  If the treatment does not reach CR/CRi/CRh after two courses, the patient is discharged.
  Consolidation therapy:
  1. intermediate-dose Ara-C (ID-Ara-C): 2 cycles are used. Ara-C 1 g/m2/q12h on days 1, 3, and 5 (for patients aged 60-70 years) or Ara-C 500 mg/m2/q12h on days 1, 3, and 5 (for patients aged 70 years or older)
  Maintenance therapy:
  VA : 6 courses
  Interventions: Drug: Venetoclax; Drug: cytarabine; Drug: azacitidine; Drug: Homoharringtonine

INTERVENTIONS:
Drug: daunorubicin — Used in combination with cytarabine and venetoclax for induction therapy in DAV.
  Arms: DAV/IAV
Drug: Venetoclax — Used in combination with cytarabine and daunorubicin for induction therapy in DAV.
Drug: cytarabine — Used in combination with venetoclax and daunorubicin for induction therapy in DAV or used by intermediate does for consolidation therapy.
Drug: azacitidine — Used in combination with venetoclax for maintenance therapy.
Drug: Homoharringtonine — Used in combination with cytarabine and venetoclax for induction therapy in HAV.
  Arms: HAV
Drug: Idarubicin — Used in combination with cytarabine and venetoclax for induction therapy in IAV.
  Arms: DAV/IAV

SUMMARY:
Acute myeloid leukemia (AML) represents the most prevalent leukemia type in China. Elderly patients (≥60 years old) have a high incidence rate, accounting for over half of all AML patients, with a median age of onset approximately 68 years. Elderly AML patients have a poor prognosis and are often accompanied with multiple high-risk factors.The 5-year overall survival (OS) is only 3-8%.

Before the advent of new targeted drugs, for elderly patients with newly diagnosed AML who were suitable for intensive chemotherapy, the most commonly used chemotherapy regimen remained the classic "3 + 7" regimen. However, the complete remission (CR) rate after induction was approximately 40-60%. The majority of elderly patients were not eligible for allogeneic hematopoietic stem cell transplantation, resulting in a relatively poor long-term survival for elderly AML patients . With the emergence of new targeted drugs, clinical studies both domestically and internationally have demonstrated that the combination of various targeted drugs and demethylating agents has achieved favorable efficacy in elderly/unsuitable for intensive chemotherapy patients with newly diagnosed AML, prolonging their survival. Previously, we initiated a multicenter, prospective, randomized controlled clinical study (registration number: NCT06066242). The aim was to explore the optimal induction regimen for elderly fit patients with newly diagnosed AML. Preliminary data revealed that the regimen of daunorubicin (DNR) or idarubicin (IDA) combined with cytarabine (Ara - C, DA/IA) + venetoclax (Ven, DAV/IAV) had a higher induction remission rate (77.3% )than the DA/IA "3 + 7" and Ven + azacitidine (AZA) regimens (45% - 59%). However, compared to the induction remission rate of young adult patients with newly diagnosed AML (> 85%), further improvement is still required.

Previous research data show that HHT enhances the inhibitory effect of Ara-c on DNA synthesis in tumor cells by influencing cell cycle regulation. The combination of HHT and Ven can jointly affect the apoptotic pathway and enhance cell apoptosis.

Therefore, this study intends to establish a prospective, randomized controlled clinical trial to compare the induction remission rates of the HHT + Ara-c + Ven (HAV) regimen with the DAV/IAV regimen, which,based on previous data, had the highest induction remission rate .

DETAILED DESCRIPTION:
This study is a multicenter, prospective, randomized, and controlled clinical trial, which intends to enroll elderly patients diagnosed with AML in accordance with the WHO (2022) or ICC standards and are suitable for intensive chemotherapy. For patients meeting the inclusion and not meeting the exclusion criteria, they will be randomly grouped and respectively receive induction therapy with either DAV/IAV (2 + 5) or HAV regimens. Patients achieving CR/CRi/CRh after induction treatment will undergo consolidation with the intermediate-dose cytarabine regimen for two courses.After completing the induction and consolidation therapy, maintenance therapy with the VA regimen for six courses will be administered; subsequently, follow-up will be conducted. Patients in the high-risk group and those with non-negative MRD are recommended to undergo allogeneic hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Conforming to the diagnostic criteria of AML or MDS/AML by WHO (2022) or ICC.
2. Age ≥ 60 years and ≤ 75 years, regardless of gender.
3. The performance status assessment of the Eastern Cooperative Oncology Group (ECOG-PS) is 0 - 2.
4. Meeting the requirements of the following laboratory examination indicators (performed within 7 days before treatment):

1) Total bilirubin ≤ 1.5 times the upper limit of normal for the same age group; 2) AST and ALT ≤ 2.5 times the upper limit of normal for the same age group; 3) Serum creatinine < 2 times the upper limit of normal for the same age group; 4) Cardiac enzymes < 2 times the upper limit of normal for the same age group; 5) The cardiac ejection fraction determined by echocardiography (ECHO) > 50%. The informed consent form must be signed before the initiation of all specific research procedures. It should be signed by the patient himself/herself or an immediate family member. Considering the patient's condition, if the patient's signature is not conducive to the treatment of the disease, the informed consent form should be signed by the legal guardian or an immediate family member of the patient.

Exclusion Criteria:

1. Acute promyelocytic leukemia accompanied by the PML-RARA fusion gene
2. Acute myeloid leukemia accompanied by the RUNX1-RUNX1T1 or CBFB-MYH11 fusion gene
3. Acute myeloid leukemia accompanied by the BCR-ABL fusion gene
4. Retreated patients (referring to those who have previously undergone induction chemotherapy but can receive hydroxyurea for cytoreduction).
5. Patients concurrently suffering from malignant tumors in other organs (requiring treatment).
6. Active cardiac diseases, defined as one or more of the following:

1) Uncontrolled or symptomatic angina pectoris history; 2) Myocardial infarction less than 6 months from the time of enrollment in the study; 3) History of arrhythmias requiring drug treatment or with severe clinical symptoms; 4) Uncontrolled or symptomatic congestive heart failure (> NYHA Grade 2);

7. Severe infectious diseases (untreated tuberculosis, pulmonary aspergillosis).

8. Those considered ineligible for enrollment by the researcher.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Up to approximately 1 years after the date of the last enrolled participants
  It is defined as the time from the start of randomization to the occurrence of induction failure or disease progression or death from any cause (whichever occurs first)

SECONDARY OUTCOMES:
Complete remission (CR) rate or complete remission with partial hematologic recovery (CRh) rate or complete remission with incomplete hematologic recovery (CRi) rate | Up to approximately eight weeks afer induction therapy
  Proportion of patients with CR, CRh or CRi
Undectable Minimal residual disease (MRD) by flow cytometry compelete remission rates after induction | Up to approximately eight weeks afer induction therapy
  Among those who have achieved CR/CRh/CRi after induction, proportion of patients who is undectable MRD by flow cytometry
Undectable Minimal residual disease (MRD) by flow cytometry complete remission rates in the whole treatment | up to 1 years after the date of the last enrolled participants
  Among those who have achieved CR/CRh/CRi in the whole treatment, proportion of patients who is undectable MRD by flow cytometry
Relapse-free Survival (RFS) | Up to approximately 1 years after the date of the last enrolled participants
  It is defined as the time from the start of achieving remission to disease progression, death from any cause or the last follow-up.
30-day postinduction mortality | Up to approximately 30 days
  It is defined as death from any cause within 30 days after the start of induction.
60-day postinduction mortality | Up to approximately 60 days
  It is defined as death from any cause within 60 days after the start of induction.
overall survival | up to 1 years after the date of the last enrolled participants
  The interval from the date of enrollment to the date of death or the date of last follow-up, whichever occurred first.

CONTACTS AND LOCATIONS:
Locations (1):
- Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No